CLINICAL TRIAL: NCT01523236
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multi-Site Study to Compare the Clinical Equivalence of Mometasone Furoate Anhydrous, 50 Mcg/Actuation Nasal Spray (Teva Pharmaceuticals USA) Compared to Nasonex® (Mometasone Furoate Monohydrate) 50 Mcg/Actuation Nasal Spray (Schering) in the Relief of the Signs and Symptoms of Seasonal Allergic Rhinitis
Brief Title: Clinical Equivalence Study of Mometasone Nasal Spray, 50 Mcg/Actuation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 70936005
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Allergic Rhinitis; Bioequivalence
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Investigational Test Product (Experimental): Mometasone furoate anhydrous 50 mcg/actuation Nasal Spray (Teva)
  Interventions: Drug: Mometasone furoate
- Reference Listed Drug (Active Comparator): Nasonex® (mometasone furoate monohydrate) 50 mcg/actuation Nasal Spray (Schering)
  Interventions: Drug: Nasonex®
- Placebo (Placebo Comparator): Saline Placebo Nasal Spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone furoate — 50 mcg/actuation Nasal Spray
  Arms: Investigational Test Product
Drug: Nasonex® — 50 mcg/actuation Nasal Spray
  Other Names: Mometasone furoate (generic name)
  Arms: Reference Listed Drug
Drug: Placebo — Nasal Spray
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the clinical equivalence of the test formulation of mometasone furoate anhydrous 50 mcg/actuation nasal spray (manufactured by Teva Pharmaceutical Industries, Ltd. and distributed by Teva Pharmaceuticals USA) to the marketed formulation Nasonex® (mometasone furoate monohydrate) nasal spray, 50 mcg/actuation (Schering) in patients with seasonal allergic rhinitis.

In addition, the efficacy of both the test and reference nasal sprays will be compared to a placebo nasal spray and safety will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female 12 years or age or older.
* Signed informed consent form, which meets all criteria of current FDA regulations. For patients under the age of majority in the state the study is being conducted (18 years in most states) the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form that will be written in such a way as to be understandable to a child.
* If female and of child-bearing potential, have a negative urine pregnancy test and is prepared to abstain from sexual intercourse or use a reliable method of contraception during the study. In order for hormonal birth control to be considered a reliable method the patient must have been on their regimen for at least 28 days.
* Documented positive allergic skin test, performed within the previous 12 months, to one or more of the allergens in season at the time the study is being conducted.
* A minimum of two years of previous history of seasonal allergic rhinitis to the pollen/allergen in season at the time the study is being conducted.
* A score of at least 6 on the reflective Total Nasal Symptom Score (rTNSS) and a minimum score of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms. The patient must meet these minimum requirements prior to being entered into the placebo lead-in period and also prior to being enrolled in the randomized, active treatment period of the study.

Exclusion Criteria:

* Under 12 years of age.
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* Negative or lack of documented skin allergen test (performed within the previous 12 months) to at least one of the allergens in season at the time the study is being conducted. The results of all positive skin allergen test results should be reported.
* Patients who suffer from chronic signs and symptoms of perennial allergic rhinitis (PAR) should be excluded from the study unless the Investigator assesses that the patient's current signs and symptoms are a clear exacerbation of Seasonal Allergic Rhinitis (SAR) rather than chronic PAR.
* Patients who suffer only from perennial allergic rhinitis of seasonal allergic rhinitis to a different allergen than that in season at the time the study in conducted.
* Previous history of less that 2 years of seasonal allergic rhinitis to the pollen/allergen in season at the time the study is being conducted.
* A total score of less than 6 on the reflective Total Nasal Symptom Score (rTNSS) or a score less than 2 for "nasal congestion" or a score less than 2 for all 3 remaining symptoms. Any patient who meets the minimum rTNSS requirements at the start of the placebo lead-in period but no longer meets the requirements prior to the randomized active treatment period of the study cannot continue in the active treatment period.
* History of asthma over the previous two years that required chronic therapy. Occasional acute or mild exercise induced asthma will be allowable on the condition that the treatment of the attacks is restricted to beta-agonists only.
* Patients with nasal conditions, including infectious rhinitis, rhinitis medicamentosa, or atrophic rhinitis.
* Clinically significant nasal deformity (e.g. significantly deformed septum, nasal polyps or ulcers) or any recent nasal surgery or trauma that has not completely healed.
* Sinus infection within the previous 30 days or history of re-occurring sinus infections.
* Patient has started immunotherapy (including topical or desensitization therapy) or changed their dose of immunotherapy within 30 days of the first placebo lead-in dose, or is likely to have to start immunotherapy or change their current dose during the study.
* Treatment for oral Candidiasis within 30 days of starting the study or a current oral Candidiasis infection.
* Upper respiratory tract infection within the previous 30 days.
* Patients with a history of tuberculosis.
* Patients with the presence of glaucoma, cataracts, ocular herpes simplex, conjunctivitis, or other eye infection not related to the diagnosis of SAR within 14 days of enrollment.
* The patient has had recent exposure (30 days) or was at risk of being exposed to chicken pox or measles.
* Patients with any untreated fungal, bacterial, or systemic viral infections within the previous 30 days.
* Use of any ophthalmic steroids within 14 days or nasal, inhaled, or systemic steroids within 30 days of the study start. Super or high potency topical steroids should not be used during the study. The use of low potency topical corticosteroids will be allowed. The use of hormonal contraceptives or hormone replacement therapy is allowed, on the condition that the patient has been on a stable dosing regime for at least 28 days prior to the start of the study and remains on the same dosing regimen during the study.
* Use of intranasal or systemic second-generation anti-histamines within 10 days of enrollment.
* Use of intranasal cromolyn within 14 days of enrollment.
* Use of intranasal or systemic first-generation anti-histamines, leukotriene receptor antagonists or other nasal decongestants within 3 days of enrollment.
* Use of any tricyclic anti-depressant within 30 days of enrollment.
* Patients with attention-deficit disorder being treated with methylphenidate containing products that have not been on a stable dosing regimen for at least 30 previous days and who cannot remain on the same dosing regime throughout the study.
* Desensitization therapy to the seasonal allergen that is causing the patient's allergic rhinitis within the previous 6 months.
* Previous SAR and/or PAR that has proven unresponsive to steroid therapy.
* Any known hypersensitivity to mometasone, other steroids, or any of the components of the study nasal spray.
* Significant history of current evidence of chronic infectious disease, system disorder, organ disorder, or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participating or could jeopardize the integrity of the study evaluations.
* Receipt of any drug as part of a research study within 30 days prior to the first placebo lead-in dose.
* Planned travel outside of the local area for more than 2 consecutive days or 3 days in total, during the patient's participation in the study.
* Previous participation in this study.
* The patient has a history or non-compliance with medication regiments or treatment protocols in previous clinical studies.
* The patient is a member of the investigational study staff or a member of the family of the investigational study staff.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline for mean reflective Total Nasal Symptom Score (rTNSS) | 2 week treatment period
  The statistical analysis for both clinical equivalence and superiority of the active treatments over placebo will involve Analysis of Covariance (ANCOVA).
  The Per-Protocol Population (PPP) will be used for the primary analysis of bioequivalence.
  The Intent-to-Treat Population (ITT) will be used for the primary analysis of superiority.

SECONDARY OUTCOMES:
Mean Change from Baseline in the mean Instantaneous Total Nasal Symptom Score (iTNSS) | 2 week treatment period
  Mean values will be presented for the secondary efficacy variable. Statistical analysis will be performed by ANCOVA.